CLINICAL TRIAL: NCT02472210
Title: A Study of the Utility of Botulinum Toxin Type A for Pain in Advanced Parkinson's Disease Double Blind Placebo Control Crossover Pilot Study
Brief Title: The Use of Botox in Advanced Parkinson's Patients Experiencing Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Susan Fox, Neurologist, Movement Disorders Clinic, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14-7474
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline IM Injection
  Interventions: Drug: Botulinum Toxin
- Onabotulinum Toxin A (Active Comparator): IM Injection
  Interventions: Drug: Botulinum Toxin

INTERVENTIONS:
Drug: Botulinum Toxin — An individualized dose will be injected in the painful limbs: up to 200 units in the upper limbs or up to 300 units in the lower limbs according to the average doses that subjects with PD pain in the limbs received in our clinic, as per our retrospective study. Each injection will contain 25 Units of Botulinum Toxin this way the number of injections will be from 1 to 8 for the upper limbs and from 1 to 12 in the lower limbs. The pattern of injections will be decided by the study investigator according to the localization. The involved muscles will be targeted using EMG guidance. of pain and will be the same at visit 2 and 3.
  Other Names: Botox

SUMMARY:
Most Parkinsonism related pain can be assigned to one or more of five categories: musculoskeletal pain, neuritic or radicular pain, dystonia associated pain, primary or central pain, and akathitic discomfort. In PD pain tends to affect the side of the body that was initially, or more severe affected by the motor symptoms. Botulinum toxins are an effective treatment modality for a growing number of neurological conditions. They have been studied for a variety of conditions associated with PD including dystonia, jaw tremor, apraxia of eyelid opening, camptocormia, dyskinesias, freezing of gait, sialhorrea, overactive bladder and constipation. There are no studies for the use of Botulinum Toxin for pain in PD. The investigators will perform a double-blind, randomized cross-over study evaluating the efficacy and safety of an individual pattern of BTXA injections targeted at painful muscles vs. placebo injection.

DETAILED DESCRIPTION:
The investigators will perform a double-blind, randomized cross-over study evaluating the efficacy and safety of an individual pattern of BTXA injections targeted at painful muscles vs. placebo injection. Primary outcome will be a measure of global pain as perceived by the participants. To assess this endpoint the investigators will use:1.

change in pain on a Numeric Rating Scale (NRS) by telephone between BTXA and placebo injections at 4 week post injection and 2.change in Visual Analogue Scale (Edmonton Symptom Assessment System: Numerical Scale) at study visits.

Secondary outcomes will be the percentage of responders, Physician rated Clinical Global Impression (CGI), Unified Parkinson Disease Rating Scale (MDS-UPDRS) on medication, quality of life by Parkinson Disease Questionnaire (PDQ-39) and adverse events as assessed at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced PD (Hoehn and Yahr 3-5) and painful limbs not responding to antiparkinsonian agents sufficiently.
* BTXA treatment naÃ-ve patients or not received any within last 12 months (including other indications).
* Stable PD and pain medications for at least 30 days
* Competence to self-report pain severity in a Visual Analogue Scale (VAS)

Exclusion Criteria:

* Subjects with a primary cause of pain unrelated with PD and associated with another medical condition e.g. severe arthritis
* Subjects that because of the severity or refractory pain are under an unfixed analgesic schedule
* Subjects unable to self- report pain severity in a VAS
* Subjects undergoing acute infections or other acute intercurrences.
* Any contraindication to receiving BTXA injections:

  1. Subjects who are hypersensitive to any BTXA or to any ingredient in the formulation or component of the container (Clostridium Botulinum toxin type A neurotoxin complex 900 kD, Human Serum Albumin and Sodium Chloride).
  2. The presence of infection at the proposed injection site(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change of patient rated pain on NRS scale | 3 months
  1. change in pain on a Numeric Rating Scale (NRS) by telephone between BTXA and placebo injections at 4 week post injection and
  2. change in Visual Analogue Scale (Edmonton Symptom Assessment System: Numerical Scale) at study visits.